CLINICAL TRIAL: NCT01557764
Title: A Phase II Study of Lapatinib in Combination With Trastuzumab in Metastatic HER2 Non-amplified But HER2 Mutant Breast Cancer
Brief Title: Lapatinib With Trastuzumab in Treating Patients With HER2-Negative/HER2 Mutant Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201206025
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor and monoclonal antibody) (Experimental): Patients receive lapatinib PO QD on days 1-21 and trastuzumab IV over 90 minutes on day 1 of a 21-day cycle. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Biological: trastuzumab

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016, GW-572016, GW2016, Lapatinib, Tykerb
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2, Herceptin, MOAB HER2, MOAB HER2, monoclonal antibody c-erb-2, monoclonal antibody HER2

SUMMARY:
This phase II trial studies the effectiveness of lapatinib ditosylate (lapatinib) together with trastuzumab in treating patients with HER2-negative breast cancer that carries HER2 gene mutations. Lapatinib may kill tumor cells by blocking some of the enzymes needed for cell division and growth. Trastuzumab, a monoclonal antibody, may block the ability of tumor cells to grow and spread. Giving lapatinib together with trastuzumab may provide a more effective treatment for patients with this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed metastatic breast cancer
* The breast cancer has been tested negative for HER2 (0 or 1+ by immunohistochemistry [IHC] or non-amplified by fluorescence in-situ hybridization [FISH])
* Patient may have measurable or evaluable disease
* If given prior radiotherapy and/or prior chemotherapy, the patient must have completed radiation therapy and be at least 1 week from the last chemotherapy administration, with adequate recovery of bone marrow and organ functions, before starting lapatinib or trastuzumab

  * Note that the HER2 sequencing analysis can be performed while patient is receiving other systemic therapies so the results could be used to determine whether the patient is eligible to receive lapatinib and trastuzumab when disease progresses from current therapy
* Patient must have had at least one lines of systemic therapy for metastatic breast cancer
* Patient must have disease that progressed on his/her most recent treatment regimen
* Patient must be > 18 years of age.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) unless due to Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 3.0 x IULN with/without liver metastases
* Creatinine =< 1.5 x IULN
* Patient must have a left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (ILLN) to be eligible for study treatment; to avoid the cost of screening, patients with known recent LVEF < LLN or symptoms of congestive heart failure are not eligible for registration
* Women of childbearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* Patient (or legally authorized representative if applicable) must be able to understand and willing to sign an institutional review board (IRB) approved written informed consent document
* Patients with known treated brain metastasis are eligible, but must have received radiation and be off steroids and stable for 3 months
* Patients meeting all inclusion criteria listed above and exclusion criteria will be registered to undergo HER2 mutation analysis; only patients with mutations in HER2 either in the primary or metastatic tumor are eligible for study therapy with lapatinib and trastuzumab; those without mutations in HER2 are not eligible for study drug therapy; information and tissue collected from patients without HER2 mutations will be used for molecular epidemiology studies of HER2 negative breast cancer

Exclusion Criteria:

* Patient must not be receiving any other investigational agents
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not have acute or currently active/requiring antiviral therapy hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment)
* Patient must not be pregnant and/or breastfeeding
* Patient must not have a history of significant cardiac disease, cardiac risk factors, or uncontrolled arrhythmias
* Patient must not have symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Overall clinical benefit rate (CBR; CD + PR + SD) of lapatinib and trastuzumab in patients with breast cancer that carry HER2 mutations | 6 months
  Responses assessed using RECIST guidelines version 1.1; duration of SD must be >= 6 months; CBR and its 80% confidence interval will be calculated.

SECONDARY OUTCOMES:
PFS of patients treated with lapatinib and trastuzumab | 2 years
  Assessed using RECIST guidelines version 1.1
Correlation of HER2 mutation with histology subtype (invasive lobular vs. invasive ductal cancer) | Baseline
Correlation of HER2 mutation with tumor grade (1-2 vs. 3) | Baseline
Correlation of HER2 mutation with tumor staging at initial diagnosis (I vs. II or III vs. IV) | Baseline
Correlation of HER2 mutation with disease free survival | 2 years
Occurrence of HER2 mutation in paired primary and metastatic sites | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu